CLINICAL TRIAL: NCT04959656
Title: Based on a Small Sample Deep Learning Multi-modal Image-assisted Diagnosis Model of Cervical Spine Tumors Clinical Application Research
Brief Title: Multimodal Imaging-assisted Diagnosis Model for Cervical Spine Tumors
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2020255
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Spine Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- X-ray: This study completed the manual labeling of preoperative multi-modal images of cervical spine structures and tumor lesions. On the normal cervical spine, six target areas were labeled: cervical spinal cord (MRI), cervical spine alignment (MRI), cervical intervertebral discs ( MRI), cervical spinal canal area (MRI), cervical cobb angle (X-ray) and cervical posterior longitudinal ligament ossification (CT). For cervical tumor lesions, complete MR and CT as well as orthopedic, axial and coronal positions. The label on the lateral X-ray image.
- CT: This study completed the manual labeling of preoperative multi-modal images of cervical spine structures and tumor lesions. On the normal cervical spine, six target areas were labeled: cervical spinal cord (MRI), cervical spine alignment (MRI), cervical intervertebral discs ( MRI), cervical spinal canal area (MRI), cervical cobb angle (X-ray) and cervical posterior longitudinal ligament ossification (CT). For cervical tumor lesions, complete MR and CT as well as orthopedic, axial and coronal positions. The label on the lateral X-ray image.
- MRI: This study completed the manual labeling of preoperative multi-modal images of cervical spine structures and tumor lesions. On the normal cervical spine, six target areas were labeled: cervical spinal cord (MRI), cervical spine alignment (MRI), cervical intervertebral discs ( MRI), cervical spinal canal area (MRI), cervical cobb angle (X-ray) and cervical posterior longitudinal ligament ossification (CT). For cervical tumor lesions, complete MR and CT as well as orthopedic, axial and coronal positions. The label on the lateral X-ray image.

SUMMARY:
Cervical spine tumor is a small sample of tumor disease with low incidence, great harm, and complex anatomical structure. It is very difficult to identify and classify benign and malignant cervical spine tumors clinically.

The deep learning model we constructed in the early stage has a higher accuracy rate for the image diagnosis of cervical spondylosis with a large number of cases, and a better clinical application effect, but the accuracy rate for cervical spine tumors with a small number of cases is lower. The reason may be the amount of data. With limited tasks, the traditional deep learning model is difficult to play an effective role.

Based on this, we propose to build a small sample-oriented deep learning model to assist clinicians in the diagnosis of cervical spine tumors with multimodal images, and to evaluate the benign and malignant tumors.

DETAILED DESCRIPTION:
Cervical spine tumor is a small-sample tumor disease with low incidence, great harm, and complex anatomical structure. It is very difficult to identify and classify benign and malignant cervical spine tumors clinically. The deep learning model we constructed in the early stage is suitable for the large number of cases. The imaging diagnosis of cervical spondylosis has a high accuracy rate and a good clinical application effect, but the accuracy rate is low for cervical spine tumors with a small number of cases. The reason may be that for tasks with limited amount of data, the traditional deep learning model is difficult to play an effective role. Based on this, we propose to construct a small sample-oriented deep learning model to assist clinicians in the diagnosis of cervical spine tumors in multi-modal imaging, and to evaluate the benign and malignant tumors. This research will not only improve the efficiency and efficiency of cervical spine tumor imaging diagnosis. Accuracy, to guide clinical personalized treatment, will also provide a basis for the clinical application of deep learning in the field of small samples, which has important clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old, about 300 males and females; in the orthopedics outpatient and emergency department of our hospital, the imaging scans (X-ray, CT, MR) showed no obvious abnormalities.

Exclusion Criteria:

* have had surgery before acquiring the images, Those who have cervical spine fractures, deformities, infections, etc. who cannot cooperate with imaging examinations, and those who have not signed the informed consent. The normal control group" includes about 600 patients with normal or slightly degenerated cervical spine, as a standard for training computers to recognize cervical spine structures Images and control images for detecting tumor lesions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion criteria: clinically suspected cervical spine tumors, multi-modality (X-ray, CT, MR) imaging, followed by needle biopsy or surgery to confirm the tumor, and pathology report. Exclusion criteria: surgery or radiotherapy before imaging, cervical spine Those who have fractures, deformities, infections, etc. who cannot cooperate with imaging examinations, and those who have not signed an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
tumor detection | 2022-2023
  On the basis of the cervical spine structure, it is the modeling of the tumor. The model based on weakly supervised learning recognizes the morphological features such as the size of the tumor lesion, and uses the fast-adapted meta-learning method to achieve a fast model under a small amount of training. Optimize, and finally evaluate the benignity, borderline and malignant probability of the tumor and use it as an output.

SECONDARY OUTCOMES:
cervical spine detection | 2022-2023
  Taking the postoperative pathology report of cancer patients as the audit standard, testing the sensitivity and accuracy of the model, and integrating it into a complete deep learning model.

CONTACTS AND LOCATIONS:
Overall Officials: hanqiang ouyang, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No